CLINICAL TRIAL: NCT01986322
Title: Phase 2 Study of Immunogenicity and Safety of DPT/HB/Hib (Bio Farma) Vaccine Compared to DTP/HB (Bio Farma) Vaccine Given Simultaneously With Hib (Registered) Vaccine in Indonesian Infants
Brief Title: Immunogenicity and Safety of DTP/HB/Hib (Bio Farma)Compared to DTP/HB Given Simultaneously With Hib(Registered)Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Penta 0211
Record Dates: First submitted 2013-10-30; First posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: DTP/HB/Hib vaccine; Immunogenicity; Infants; Safety
MeSH Terms: interventions — HibTITER protein, Haemophilus influenzae

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DTP/HB/Hib vaccine (Experimental): Group A will receive DTP/HB/Hib combination vaccine at 6-11, 10-15 and 14-19 weeks of age.
  DTP/HB/Hib component:
  Purified diphteria toxoid Purified tetanus toxoid Inactivated Bordetella pertussis HbsAg PRP-TT Aluminum phosphate Natrium Chloride Thimerosal
  Interventions: Biological: DTP/HB/Hib vaccine
- DTP/HB and Hib vaccine (Active Comparator): Group B will receive DTP/HB and Hib Vaccines separately at 6-11,10-15, 14-19 weeks of age
  DTP/HB component:
  Purified diphteria toxoid Purified tetanus toxoid Inactivated Bordetella pertussis rHbsAg Aluminum phosphate Natrium Chloride Thimerosal
  Hib component:
  Purified Haemophilus influenzae type b polysaccharide 10 mcg
  Interventions: Biological: DTP/HB and Hib vaccine

INTERVENTIONS:
Biological: DTP/HB/Hib vaccine — Dosage equal to 0.5 mL administered intramuscularly
  Other Names: Pentavalent
  Arms: DTP/HB/Hib vaccine
Biological: DTP/HB and Hib vaccine — Dosage equal to 0.5 mL administered intramuscularly
  Arms: DTP/HB and Hib vaccine

SUMMARY:
The main objective of this study was to evaluate the protectivity and safety of DTP/HB/Hib (Bio Farma) vaccine compared to DTP/HB and Hib vaccine given simultaneously.

DETAILED DESCRIPTION:
This trial was randomized, single blind, prospective intervention study. Total 220 subject (6-11 weeks of ages) followed this trial, divided into 2 groups, each group consists of 110 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Infant 6-11 week of age
* Infant born after 37-42 week of pregnancy
* Infant weighing more than 2.5 kg at birth
* Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form
* Parents commit themselves to comply with the indication of the investigator and with the schedule of the trial
* Mother at least graduate from elementary school
* Received Hepatitis B vaccine (Bio Farma) at birth

Exclusion Criteria:

* Child concomitantly enroll or schedule to be enroll in another trial
* Evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature >=37.5 Celsius on Day 0)
* Known history of allergy to any component of the vaccine component (e.g.formaldehyde)
* History of uncontrolled coagulopathy or blood disorder contraindicating intramuscular injection
* Known history of congenital or acquired immunodeficiency (including HIV infection)
* Child who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulin, blood derived product or long term corticotherapy (>2 weeks)
* Other vaccination within the 7 days prior to inclusion with the exception of BCG and poliomyelitis
* Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objective
* Infant with a known history of diphteria, tetanus, pertussis, Hib, Hepatitis B infection

Ages: 6 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Protectivity of DTP/HB/Hib (Bio Farma) vaccine | 4 months
  Percentage of infants with anti diphteria titer and anti tetanus titer >= 0.01 IU/ml, AntiHbs titer >=10mlIU/ml, and antiPRP-TT titer >= 0,15ug/ml 28 days after the last injection (third) in DPT/HB/Hib liquid vaccine group

SECONDARY OUTCOMES:
Antibody response to diphteria toxoid in both group | 4 months
  Serological response to diphteria toxoid: GMT, percentage of infants with titer >=0.01 IU/ml and >=0.1 IU/ml, percentage of infants with increasing antibody titer >=4 times and/or percentage of infants with transition of seronegative to seropositive.
Antibody response to Tetanus Toxoid in both group | 4 months
  Serological response to tetanus toxoid: GMT, percentage of infants with titer >=0.01 IU/ml and >=0.1 IU/ml, percentage of infants with increasing antibody titer >=4 times and/or percentage of infants with transition of seronegative to seropositive
Antibody response to Pertussis component in both group | 4 months
  Serological response to the pertussis component (agglutinins): GMT,percentage of infants with titre >=40, >=80,>=160 and >=320 (1/dil.), percentage of infants with increasing antibody titer >=4 times.
Antibody response to Hepatitis B in both group | 4 months
  Serological response to Hepatitis B: Geometric mean of anti-HBs, percentage of infants with titer >=10mlIU/ml, percentage of infants with increasing antibody titer >=4 times and/ or percentage of infants with transition of seronegative to seropositive.
Antibody response to PRP-T in both group | 4 months
  Serological response to Hib/PRP: GMT, percentage of infants with titre >=1ug/ml and >=0.15ug/ml, percentage of infants with increasing antibody titer >=4 times and/or percentage of infants with transition of seronegative to seropositive
Incidence rate of adverse event of DTP/Hepatitis B/Hib vaccine (Bio Farma) | 30 minutes, 72 hours, 28 days after immunization
  Local and systemic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Kusnandi Rusmil, PhD, Principal Investigator — Faculty of Medicine UNPAD
Locations (3):
- Indonesia (3):
  - Garuda Primary Health Center, Bandung, West Java
  - Ibrahim Adji Primary Health Care Center, Bandung, West Java
  - Puter Primary Health Center, Bandung, West Java